CLINICAL TRIAL: NCT05731375
Title: Mitochondrial dysfUnction: a Key Player in Doxorubicin-induced Skeletal and Cardiac muscLE Damage
Acronym: MUSCLE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Julius Clinical (Industry)
Responsible Party: Principal Investigator, Dr. Anne May, Prof. Dr., UMC Utrecht
Other Study IDs: NL83538.041
Record Dates: First submitted 2023-01-25; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Doxorubicin Induced Cardiomyopathy; Chemotherapeutic Toxicity; B-cell Lymphoma; T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Patients with large B-cell lymphoma or T-cell lymphoma scheduled for 6 full-dose cycles of 1st line immunochemotherapy with (R-)CHOP
  Interventions: Diagnostic Test: 31-MRS at 7 Tesla (T)

INTERVENTIONS:
Diagnostic Test: 31-MRS at 7 Tesla (T) — 31-MRS imaging at 7T to evaluate mitochondrial function in skeletal and cardiac muscles.

SUMMARY:
The goal of this observational study is to demonstrate the ability of using non-invasive Phosphorus (31P) Magnetic Resonance Spectroscopy (MRS) to monitor changes of in-vivo markers of mitochondrial function in skeletal and cardiac muscles in muscles in large B- or T-cell lymphoma patients during treatment with (R-)CHOP. The main question it aims to answer is:

• Can 31P-MRS be used to monitor changes of in vivo markers of mitochondrial function in skeletal and cardiac muscles in large B- or T-cell lymphoma patients during treatment with (R-)CHOP?

To be able to answer this main question, participants will undergo 31P-MRS imaging of the calf muscles and of the heart 3 times during the study period.

DETAILED DESCRIPTION:
Rationale: Patients with large B-cell lymphoma or T-cell lymphoma are often treated with (R-)CHOP chemotherapy with the intent to cure the disease, but this treatment can also lead to serious toxicities, which may last for many years. (R-)CHOP contains doxorubicin, which has detrimental effects on skeletal and cardiac muscles. Loss of skeletal muscle mass is associated with treatment modifications (i.e., dose delay/reduction/discontinuation), increased levels of fatigue, decreased quality of life (QoL) and shorter survival. Cardiomyopathy might lead to chronic heart failure in the long-term, which negatively affects prognosis as well. Preclinical studies investigating underlying mechanisms of these detrimental effects suggest that mitochondrial dysfunction plays a key role. However, human data is lacking due to the need of invasive repeated muscle biopsies. Phosphorus (31P) Magnetic Resonance Spectroscopy (MRS) is an innovative, non-invasive technique, which enables repeated measures of skeletal and cardiac muscle mitochondrial energy metabolism.

Hypothesis:

In this study the investigators hypothesize that patients with large B-cell lymphoma or T-cell lymphoma treated with (R-)CHOP will show decreased mitochondrial function in skeletal and cardiac muscle tissue following chemotherapy treatment.

Objective:

To demonstrate the ability of using non-invasive 31P-MRS to monitor changes of in vivo markers of mitochondrial function in skeletal and cardiac muscles (i.e., skeletal muscle PCr recovery rate constant and cardiac PCr/ATP ratio) in patients with large B-cell lymphoma or T-cell lymphoma during treatment with (R-)CHOP. Furthermore, the investigators will assess the feasibility of undergoing the study measurements for patients with large B-cell lymphoma or T-cell lymphoma during intensive (R-)CHOP treatment and explore the association between changes in in vivo measured mitochondrial function in skeletal and cardiac muscle tissue and changes in muscle mass, physical fitness, muscle strength, physical activity levels measured by Fitbit, chemotherapy completion rate and patient-reported outcomes, including physical activity, fatigue and quality of life.

Study design: Cohort study.

Study population: Patients with large B-cell lymphoma or T-cell lymphoma scheduled for 6 full-dose cycles of 1st line immunochemotherapy with cyclophosphamide, doxorubicin, vincristine and prednisone with or without rituximab ((reversed) (R-)CHOP).

Main study parameters/endpoints:

The main study parameters are differences in skeletal muscle PCr recovery rate constant and cardiac PCr/ATP ratio. These parameters will be compared within-patients before, halfway during and after completion of chemotherapy treatment.

Nature and extent of the burden and risks associated with participation and benefit:

Included patients will visit the UMC Utrecht 3 times (i.e., before, halfway during and after completion of chemotherapy treatment). During these visits, participants will undergo 31P-MRS imaging of the calf muscles and of the heart at 7 Tesla. During the calf muscle scan, patients will be asked to perform a mild exercise challenge (i.e., dynamic plantar flexions). 7T 31P-MRS is a safe and reliable technique for subjects without contra-indications for undergoing MRI. Possible side-effects are limited to short-term vertigo and nausea. In addition, anthropometrics will be measured and small tests to evaluate muscle strength and physical performance will be performed. Participants will be asked to complete questionnaires regarding physical activity, quality of life and fatigue. Finally, patients will be asked to wear a Fitbit, provided by the study team, to objectively assess their levels of physical activity.

Subjects will not experience direct benefits by participating in this study. By the end of the study, the investigators will demonstrate the ability to non-invasively monitor skeletal and cardiac muscle mitochondrial damage using 31P-MRS, which is a pre-requisite to assess the efficacy of (non-)pharmacological interventions.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Patients with large B-cell lymphoma or T-cell lymphoma scheduled for 6 full-dose cycles of 1st line immunochemotherapy with cyclophosphamide, doxorubicin, vincristine and prednisone with or without rituximab ((reversed) (R-)CHOP).
* WHO-performance score 0-2.
* Patients with sufficient Dutch writing and reading skills.
* Written informed consent.

Exclusion Criteria:

* Contra-indications for 7T MR scanning, including patients with a non-MRI compatible pacemaker, cochlear implant or neurostimulator; patients with non-MR compatible metallic implants in their eye, spine, thorax or abdomen; patients with a non-MR compatible aneurysm clip in their brain; patients with claustrophobia, and/or severe obesity.
* Any circumstances that would impede adherence to study requirements or ability to give informed consent.
* Medical disorders affecting mitochondrial function; e.g., spinal muscular atrophy.
* (Other) relevant medical disorders; e.g., comorbidities affecting exercise tolerance.
* Being under examination for non-diagnosed disease at the time of investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at UMC Utrecht, Diakonessenhuis Utrecht and possibly other hospitals in the vincity of the UMC Utrecht. The aim is to include 12 patients with large B-cell lymphoma or T-cell lymphoma, who are scheduled to undergo (R-)CHOP treatment at any of the recruiting hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in skeletal and cardiac muscle mitochondrial function | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  Assessed through 31P-MRS imaging. Parameters include:
  * PCr recovery rate (in seconds)
  * PCr/ATP ratio

SECONDARY OUTCOMES:
Adherence rates to the study protocol | Baseline to 18 weeks.
  Measured as:
  * recruitment/retention rates
  * completion of study measurements within timeframes
Changes in physical fitness (Maximum short exercise capacity (Watt)) | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  Assessed through Steep Ramp test
Changes in hand grip strength (kg) | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  Assessed through Hand Grip Strength Test
Changes in leg strength (kg) | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  Assessed through hypothetical 1-repetition max leg press
Changes in skeletal muscle area in cm2 | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  Assessed through routine CT-scans
Changes in subjective physical activity levels (min/week moderate-to-vigorous physical activity) | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  Physical activity levels will be assessed subjectively using the Short QUestionnaire to ASsess Health-enhancing physical activity (SQUASH)
Changes in objective physical activity levels (min/week moderate-to-vigorous physical activity) | Throughout the whole study, but of particular interest are the 9th week after baseline and 18th week post-baseline
  Participants are provided with a Fitbit Inspire HR and are asked to wear these as much as possible during the whole study period. The Fitbit continuously registers the heart rate. Based on this, physical activity levels will be calculated.
Changes in health-related Quality of Life | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  Measured using the core EORTC Quality of life questionnaire (QLQ-C30). The results of the questionnaire can be used to calculate a summary score, global health status, functional subscales and symptom subscales. For the summary score, global health status and functional subscales, a higher score is a better outcome, whilst for the symptom subscales, a lower score is a better outcome. All scores range from 0 to 100.
  * Global health status
  * Summary score
  Functional scales:
  * Physical functioning
  * Role functioning
  * Emotional functioning
  * Cognitive functioning
  * Social functioning
  Symptom scales:
  * Fatigue
  * Nausea and vomiting
  * Pain
  * Dyspnoea
  * Insomnia
  * Appetite loss
  * Constipation
  * Diarrhoea
  * Financial difficulties
Changes in lymphoma specific symptoms | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  Measured using the add-on of the abovementioned EORTC QLQ-C30, which is specifically developed for non-Hodgkin lymphoma patients (EORTC QLQ-NHL-HG29). A higher score depicts worse outcomes. All scores range from 0 to 100.
Changes in fatigue | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  The EORTC provides several questionnaires to asses the quality of life of cancer patients. To assess fatigue the EORTC developed a specific fatigue questionnaire (QLQ-FA12). This questionnaire can be used to assess different dimensions of fatigue. A lower score depicts a better outcome. All scores range from 0 to 100.
  Fatigue dimensions:
  * Physical fatigue
  * Emotional fatigue
  * Cognitive fatigue
Changes in skeletal muscle end-exercise pH | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  Assessed through 31P-MRS imaging.
Changes in skeletal muscle delta PCr during recovery after exercise in mM | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  Assessed through 31P-MRS imaging.

OTHER OUTCOMES:
Changes in weight (kg) | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  As measured by investigator during study visit.
Height (cm) | Baseline, halfway (R-)CHOP treatment (+/- 9 weeks), after (R-)CHOP treatment (+/- 18 weeks)
  As measured by investigator during study visit.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Diakonessenhuis, Utrecht
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
As the data is privacy-sensitive, the investigators will publish the descriptive metadata in the data repository with a description of how a data request can be made (by sending an email to the corresponding author). In the event that peers like to reuse our data this can only be granted if the research question is in line with the original informed consent signed by the study participants. Every application therefore wille be screened for this requirement. If granted, a data usage agreement is signed by the receiving party.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data and documentation needed to reproduce findings from this study will be stored for at least 15 years.
Access Criteria: Data access can only be granted for research with a research question in line with the original informed consent signed by the study participants.